CLINICAL TRIAL: NCT07087314
Title: A Clinical Study to Evaluate the Initial Efficacy and Safety of Anti-CD38 Monoclonal Antibody (SG301) Subcutaneous Injection in Children With Frequent Relapses or Steroid-Dependent Nephrotic Syndrome
Brief Title: A Study of Anti-CD38 Monoclonal Antibody (SG301) Subcutaneous Injection in Children With Nephrotic Syndrome With Frequent Relapses or Steroid Dependence
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mao Jianhua (Other)
Responsible Party: Sponsor-Investigator, Mao Jianhua, Professor, The Children's Hospital of Zhejiang University School of Medicine
Organization: The Children's Hospital of Zhejiang University School of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSG-301 SC-204
Record Dates: First submitted 2025-07-09; First posted 2025-07-25 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Nephrotic Syndrome in Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SG301 Subcutaneous injection (Experimental): full - dose prednisone (60 mg/m²/day, up to 80 mg) for remission induction. After 3 days of negative urine protein, start SG301 Subcutaneous injection with steroid tapering. Taper prednisolone to 60 mg/m² (max 80 mg) every other day, reducing by 1/6 every 2 weeks, and stop after 3 months.
  Interventions: Drug: SG301 Subcutaneous injection

INTERVENTIONS:
Drug: SG301 Subcutaneous injection — Subcutaneous injection every weeks (QW*6),subsequently, administer it once every two weeks for a total of three times (Q2W*3). The total number of doses is nine.

SUMMARY:
This is an open - label study to evaluate the safety, pharmacokinetics, pharmacodynamics, and preliminary efficacy of SG301 Subcutaneous injection in children with frequently relapsing or steroid - dependent nephrotic syndrome.

DETAILED DESCRIPTION:
This study will recruit children aged 6 - 18 with frequently relapsing or steroid - dependent nephrotic syndrome, who have morning urine protein < 1 + or urine protein / creatinine < 0.2 g/g (<20 mg/mmol) for at least three consecutive days after steroid treatment.

The study will stratify participants into two age groups:≥6 - <12 years and≥12 - <18 years. Recruitment will start with the 12 - 18 - year - old group. After collecting sufficient safety and clinical pharmacology data to support moving to lower age groups, the 6 - 12 - year - old group will be recruited. For every 1 to 3 participants enrolled, there will be a phased data review to guide further recruitment.

The trial has three phases: screening (D - 28~D - 1), treatment (12 - week), and follow - up (40 - week). The enrolled participants will be treated with 12 mg/kg SG301 Subcutaneous injection subcutaneously. They will receive weekly injections for the first six weeks, then every two weeks for three times, totaling nine injections.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 6 - 18 years.
2. Steroid-sensitive nephrotic syndrome with frequent relapses (FRNS) or steroid dependence (SDNS).
3. Normal renal function: eGFR≥90 ml/min/1.73m².
4. After steroid treatment, morning urine protein<1 + or urine protein/creatinine<0.2 g/g (<20 mg/mmol) for ≥3 consecutive days.
5. Within 7 days before enrollment, blood tests (without growth factors or transfusions) must meet: hemoglobin>80 g/L; platelets>75×10⁹/L; neutrophils>1.5×10⁹/L.
6. Prothrombin time/INR≤1.5×ULN, unless due to anticoagulation.
7. No Tacrolimus, cyclosporine A, mycophenolate mofetil, belimumab, levamisole, azathioprine, or cyclophosphamide in prior 2 months; no rituximab or obinutuzumab in prior 6 months.

Exclusion Criteria:

1. Family history of nephrotic syndrome, chronic glomerulonephritis, or uremia.
2. Alanine aminotransferase >2×ULN or total bilirubin>2×ULN with a sustained increase for 2 weeks.
3. HBsAg or HBcAb positive with Hepatitis B virus DNA above the lower limit of normal; Hepatitis C virus antibody - positive with Hepatitis C virus RNA positive; HIV antibody - positive.
4. Chronic active infections (e.g., Epstein-Barr Virus, Cytomegalovirus, tuberculosis) that may worsen with steroids/ immunosuppressants.
5. Acute active infection (excluding onychomycosis) requiring systemic antibiotics/antivirals.
6. Secondary nephrotic syndrome (e.g.,immunoglobulin A - associated, lupus nephritis); steroid - resistant nephrotic syndrome (SRNS).
7. Other autoimmune diseases, primary immunodeficiency, or malignancy.
8. Prior anti - cluster of differentiation 38 (CD38) treatment.
9. Live/attenuated vaccine receipt or major surgery (non - diagnostic) within 4 weeks before first dose.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2028-07-09 (Estimated); Study Completion 2029-07-09 (Estimated)

PRIMARY OUTCOMES:
Incidence and rate of treatment-Emergent Adverse Events | From baseline through study completion, an average of 1 year
  Number and percentage of adverse events which are calculated by worst CTCAE grade by CTCAE 5.0
Relapse free survival rate | Average 1 year per subject
  Relapse free survival rate at 6 and 12 months

SECONDARY OUTCOMES:
Relapse frequency in times | From baseline through study completion, an average of 1 year
  Proportion of relapsed participants
Time to Relapse | From baseline through study completion, an average of 1 year
  Time to first relapse after enrollment
Serum creatinine | From baseline through study completion, an average of 1 year
  Serum creatinine(SCr), SCr in mg/dl
estimated glomerular filtration rate | From baseline through study completion, an average of 1 year
  Estimated glomerular filtration rate (eGFR), eGFR in ml/min/1.73m²
Cumulative corticosteroid dose | From baseline through study completion, an average of 1 year
  The total amount of corticosteroids used during the study period, and the total amount of corticosteroids used in the 6 months prior to enrollment
SG301 anti-drug antibodies | From baseline through study completion, an average of 1 year
  Number of subjects positive for anti-SG301 anti-drug antibodies
Neutralizing antibodies against SG301 | From baseline through study completion, an average of 1 year
  the neutralizing antibody titer of anti-SG301 anti-drug antibodies
pharmacokinetics : Ctrough | From baseline through study completion, an average of 1 year
  The trough concentration of SG301

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Henan Children's Hospital Zhengzhou Children's Hospital, Zhengzhou, Henan
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei
  - Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No